CLINICAL TRIAL: NCT00002271
Title: An Ascending, Single Oral Dose Pharmacokinetic Study of 3'-Deoxy-3'-Fluorothymidine (FLT) in Asymptomatic Human Immunodeficiency Virus (HIV)-Infected Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lederle Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 054A; 81-1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-06

CONDITIONS: HIV Infections
Keywords: Thymidine; Nucleosides; Antiviral Agents
MeSH Terms: conditions — HIV Infections | interventions — alovudine

INTERVENTIONS:
Drug: Alovudine

SUMMARY:
To characterize the pharmacokinetics of orally administered 3'-deoxy-3'-fluorothymidine (FLT), in a liquid formulation, after single doses in asymptomatic HIV-infected patients and to assess the safety and tolerance of the single oral doses of FLT.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Oral candida infection documented by morphology or by response to antifungal therapy within 2 months prior to study entry.
* Temperature > 37.8 degrees Centigrade.
* Malignancy other than cutaneous basal cell carcinoma or cervical carcinoma in situ.
* Significant chronic underlying medical illnesses which would prevent continuous participation in this clinical trial.

Concurrent Medication:

Excluded:

-

Patients with the following are excluded:

* Significant chronic underlying medical illnesses which would prevent continuous participation in this clinical trial.
* Unwilling to sign informed consent.
* Intolerant to zidovudine (AZT).
* Oral hairy leukoplakia at any time prior to study entry.

Prior Medication:

Excluded within 7 days of study entry:

* Antiretroviral drugs.
* Immunomodulators.
* Excluded within 30 days of study entry:
* Any investigational drugs.

Patients have the following:

* HIV seropositivity by licensed ELISA test, confirmed by Western Blot analysis.
* No symptoms as defined by:

  1. Normal neurological exam.
  2. Absence of the following:
* Unintentional weight loss of greater than 10 pounds or more than 10 percent of usual body weight within 2 months prior to study entry.
* Unexplained temperature > 37.8 C on more than 5 consecutive days or on more than 10 days in any 30 day period in the one month prior to expected study entry.
* Unexplained diarrhea defined by = or > 3 liquid stools per day persisting > 7 days within 2 months prior to expected study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States